CLINICAL TRIAL: NCT03060681
Title: Thoracolumbar Interfacial Plane Block for Analgesia After Spine Surgery
Brief Title: Thoracolumber Oterfacial Plane Block for Spine Surgery
Acronym: TLIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, lecturer of anesthesia, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TLIP
Record Dates: First submitted 2017-02-11; First posted 2017-02-23 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Spine Surgeries
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T group (Experimental): Ultrasound guided Bilateral TLIP Block will be performed 15 minute before the start of surgery Using 15 ml of bupivacaine 0.25 for each side.
  Interventions: Drug: Bupivacaine 0.5% injected in the thoraco-lumber inetrfacial plane block
- C group (No Intervention)

INTERVENTIONS:
Drug: Bupivacaine 0.5% injected in the thoraco-lumber inetrfacial plane block — After attaching basic monitors (ECG, SpO2, NIBP), the patient will take the prone position. Using the superficial probe of the ultrasound machine, the probe will be placed in transversally in midline position at selected level. The spinous process and interspinalis muscles will be identified. The probe was then moved laterally to identify the mulifidus muscle (MF) and the longissimus muscles (LG) where the local anesthetic will be injected. The needle will be advanced under real-time in-plane ultrasound guidance till it reaches the interface between the two muscles then a 1-2 ml of saline will be inserted to confirm needle site. 15 ml of bupivacaine 0.25 will be injected each side.
  Arms: T group

SUMMARY:
The most commonly used technique to anesthetize patients scheduled for thoracic or lumbar spine surgery is general anesthesia. Analgesic techniques vary from the use of neuraxial techniques like epidural, intrathecal, or caudal analgesia, nerve root infiltration to the use of systemic opioids, Paracetamol, non-steroidal anti-inflammatory drugs (NSAID), steroids and gabapentinoids .

In 2015, a promising regional analgesia technique was reported, that targets the dorsal, rather than ventral, rami of the thoracolumbar nerves as they pass through the paraspinal musculature, and called this a thoracolumbar interfacial plane block (TLIP).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for Spine surgery.

Exclusion Criteria:

* Spine deformities, redo surgeries, patients refusing being enrolled in the study, and patients with a bleeding tendency (INR˃ 1.4 and or Platelet count ≤ 150 X103/ µl) will be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-02-20 (Estimated); Study Completion 2018-02-20 (Estimated)

PRIMARY OUTCOMES:
postoperative morphine consumption in milligrams | for the 1st 24 hours after surgery
  morphine consumption (mg)required to keep visual anlohue scale below 4 in the 1st 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided